CLINICAL TRIAL: NCT00955461
Title: Post-Market, Randomized, Single Blind, Split-Faced Comparison of the RevLite Nd:YAG Laser System Versus a Non-Ablative, Mid Infra-red, Fractionated Type Laser System for Skin Rejuvenation
Brief Title: Comparison of the RevLite Electro-optic Q-Switched Neodymium-doped Yttrium Aluminium Garnet (EO QS Nd:YAG) Laser to a Fractionated Laser System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConBio, a Cynosure Company (Industry)
Responsible Party: Sponsor
Organization: Cynosure, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C66-07-F
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Photodamage; Irregular Pigmentation; Acne Scars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser treatment (Experimental): Split-Face Comparison of an Electro-optic Q-Switched Nd: YAG Laser to a Fractionated Laser
  Interventions: Procedure: RevLite laser treatment; Procedure: Fractionated Laser treatment

INTERVENTIONS:
Procedure: RevLite laser treatment — Electro-optic Q-Switched Nd: YAG Laser treatment
Procedure: Fractionated Laser treatment

SUMMARY:
The purpose of this study is to compare the results of treatment between the side of the face treated with the RevLite Laser and the side of the face treated with a fractionated laser system.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I-VI and Wrinkle Class I
* Between the ages of 25-65
* Evidence of bilateral dyschromia

Exclusion Criteria:

* Pregnant, lactating, or is planning to become pregnant
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* any skin pathology/condition that could interfere with evaluation or requires the use of interfering topical or systemic therapy
* coagulation disorder or currently using anti-coagulation medication (including but not limited to heavy aspirin therapy)
* any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in the study
* currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 30 days
* unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
* unreliable for the study, including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits
* Accutane within 6 months
* need to be exposed to artificial tanning devices or excessive sunlight during the trial
* prior treatment with parenteral gold therapy
* Diabetes Type 1 or 2
* does not agree to refrain from any other type of facial skin resurfacing (e.g., microdermabrasion, laser or IPL treatment, chemical peel) or injected fillers/other substances (e.g., Restylane, Botox) that might affect the treatment area for the duration of the study
* artificial tanning within 1 month
* (micro)dermabrasion within 3 months
* other laser or IPL to the face within 6 months
* chemical peel within 1 month
* injectable fillers within 3 months
* topical retinoids within 3 months
* over-the-counter anti-aging products (e.g., those containing peptides, hyaluronic acid, or agents specifically advertised as having anti-aging or age-inhibiting properties) within 1 month
* history of keloids or hypertrophic scarring
* evidence of compromised wound healing
* history of cold sores, chickenpox or shingles and unwilling to take a prophylactic course of Valtrex/acyclovir
* allergy to acyclovir

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the percentage of overall, cumulative improvement from Baseline in the appearance of wrinkles, skin tone and/or texture, pigmentation and acne scars | 3 and 6 months post final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sadick, MD, Principal Investigator — Sadick Research Group
Locations (1):
- Sadick Research Group, New York, New York, United States